CLINICAL TRIAL: NCT02089100
Title: Multicentric Phase III Trial of Superiority of Stereotactic Body Radiation Therapy in Patients With Metastatic Breast Cancer in First-line Treatment
Brief Title: Trial of Superiority of Stereotactic Body Radiation Therapy in Patients With Breast Cancer
Acronym: STEREO-SEIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00142-43; 2013/1957 (Other: CSET number)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stereotactic body radiation therapy (Experimental): The SBRT of all metastases should start in maximum 4 weeks after randomization. Beginning of systemic treatment will take place before 2 and 7 days after SBRT completion. All metastases lesions should be treated every 48h.
  Interventions: Radiation: stereotactic body radiation therapy; Radiation: Systemic treatment
- no specific treatment (Active Comparator): no specific treatment to the oligometastatic sites except for palliation (pain, compression, hemorrhage)
  Interventions: Radiation: Systemic treatment

INTERVENTIONS:
Radiation: stereotactic body radiation therapy
  Arms: stereotactic body radiation therapy
Radiation: Systemic treatment

SUMMARY:
The previous reported phase I study allows us to prospectively define the optimal total dose in different metastatic locations (88). However, several questions are still unanswered such as the adequate timing of the stereotactic body radiation therapy (SBRT) in oligometastatic disease. Indeed, there are two different oligometastatic states: "de novo", i.e. occurring at first metastatic presentation without any previous systemic therapy; and "secondary", defined as residual disease after systemic treatment.

The investigators wish to prospectively study the role of metastases SBRT with curative intent in de novo oligometastatic disease.

This clinical trial would be the first randomized study studying SBRT at onset of the metastatic disease. If this trial shows a PFS improvement, it will definitively change the standard of treatment and it will highlight SBRT as a key treatment of metastatic disease. It will confirm the oligometastasis hypothesis as well as the Simon Norton hypothesis (92).

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven breast cancer stage IV AJCC TNM
2. Age >18 years
3. WHO status</=2
4. Hormonal receptors positive breast cancer (IHC)
5. The primary tumor was treated or will be treated with curative intent (surgery and /or radiotherapy)
6. No prior treatment for metastatic relapse. It will be accepted patients which would have begun a treatment in the case where:

   1. Hormonotherapy </= 1 month
   2. Chemotherapy </= 1 cycle

   The treatment must be stopped after signature of the consent form.
7. a. Metastatic lesions out of previous radiation field;

   b. Equal or less than 5 metastatic lesions (measurable or not);

   c. In case of measurable lesions, each </=10 cm or </=500 mL
8. For liver mets:

   1. adequate liver function (liver enzyme <3N, bilirubin <30mg/dl, albumin >2.5g/dl)
   2. no underlying cirrhosis or hepatitis
   3. liver metastase size </=7cm diameter
   4. not adjacent to stomach or small bowel
9. For abdominal mets:

   a. adequate renal function with a creatinine clearance (Cockroft formula) > 60ml/min
10. Absence of any psychological, familial, sociological or geographical condition with a potential to hamper compliance with the study protocol and follow-up schedule
11. Life expectancy > 3 months
12. Affiliated to Health Insurance regimen
13. Written and signed consent form

Non-inclusion Criteria:

1. Triple negative breast cancer
2. Prior systemic treatment in metastatic setting (endocrine therapy, chemotherapy, targeted therapies, radionuclide)
3. Brain metastases
4. In spinal cord mets:

   1. More than 3 consecutive and contiguous spinal segments involved by tumor
   2. Neurological examination prior randomization > 1 week
   3. Inability to tolerate treatment (unable to lie flat)
   4. Treated with radionuclide/systemic chemotherapy within 30 days before SBRT
   5. Significant or progressive neurological deficit
   6. More than 25% spinal canal compromise
   7. Malignant epidural spinal cord compression or cauda equina syndrome
   8. Spine instability or neurological deficit resulting from bony compression of neural structures
5. Scleroderma or connective tissue disease as a contraindication to radiotherapy
6. Pregnancy or breast feeding period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2014-02; Primary Completion 2025-06 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | evaluated with a minimal follow-up of 3 years in all patients
  events: local recurrence, distant progression of the target metastases, any new metastasis, death of any cause The definition of progression is based on RECIST1.1 criteria. Progression is assessed locally, in any metastasis present at the time of randomization or in any newly diagnosed metastasis.

SECONDARY OUTCOMES:
Cumulative rate of local failure | evaluated with a minimum follow-up of 3 years in all patients.
  assessed with RECIST1.1 criteria
Overall survival | evaluated with a minimum follow-up of 3 years in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Céline BOURGIER, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France